CLINICAL TRIAL: NCT02448446
Title: The Effect of Intravitreal Ranibizumab on Visual Acuity and Hard Exudate Resolution in the Treatment of Diabetic Macular Edema With Foveal Involving Edema and Lipid Exudates
Brief Title: The Effect of Intravitreal Ranibizumab on Visual Acuity and Hard Exudate Resolution in the Treatment of Diabetic Macular Edema With Center Involved Edema and Lipid Exudates
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: South Coast Retina Center; Carson, McBeath, Boswell, Inc. (Other)
Collaborators: Genentech, Inc. (Industry); Doheny Image Reading Center (Other); The Retina Partners (Other)
Responsible Party: Principal Investigator, Julie Gasperini, M.D., Medical Doctor, South Coast Retina Center; Carson, McBeath, Boswell, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML259577
Record Dates: First submitted 2015-03-05; First posted 2015-05-19 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Macular Edema; Hard Lipid Exudates
MeSH Terms: interventions — Ranibizumab

ARMS (2):
- Diabetic macular edema treatment group (Group 1) (Active Comparator): Treatment using intravitreal ranibizumab 0.3mg based on the DRCR protocol I 4:2:7 strategy based on the presence of macular edema.
  Interventions: Drug: ranibizumab 0.3mg
- Diabetic macular edema and lipid treatment group (Group 2) (Active Comparator): Continued treatment with intravitreal ranibizumab 0.3mg until, not only the macular edema is resolved, but also until the lipid exudate is resolved.
  Interventions: Drug: ranibizumab 0.3mg

INTERVENTIONS:
Drug: ranibizumab 0.3mg — intravitreally administered
  Other Names: Lucentis

SUMMARY:
This is an open-label, Phase I/II study of intravitreally administered 0.3mg ranibizumab in subjects with diabetic macular edema and lipid exudates in the central subfield.

DETAILED DESCRIPTION:
This is an open-label, Phase I/II study of intravitreally administered 0.3mg ranibizumab in subjects with diabetic macular edema and lipid exudates in the central subfield.

Consented, enrolled subjects will receive multiple open-label intravitreal injections on 0.3mg ranibizumab administered every 30 days for 12 months per the treatment algorithm.

The patients will be randomized to 1 of 2 treatment groups. Group 1: Treatment algorithm based on the Diabetic Retinopathy Clinical Research (DRCR) protocol I 4:2:7 strategy based on the presence of macular edema.

Group 2: Continue treatment until not only the macular edema is resolved but also until the lipid exudate is resolved.

Sample size: 30 eyes Follow-up Schedule: Every 4 weeks throughout the study.

ELIGIBILITY:
Subjects will be eligible if the following criteria are met:

Inclusion Criteria

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age ≥ 18 years
* Type 1 or Type 2 Diabetes mellitus
* Best corrected ETDRS visual acuity (20/32-20/320) or letter score 78 to 24
* Diabetic macular edema on clinical examination involving the center of the macula assessed to be the main cause of visual loss
* Retinal thickness measured on spectral domain optical coherence tomography (OCT). Zeiss Cirrus: ≥290μm in women and ≥305 μm in men in the central subfield. Heidelberg Spectralis: ≥305μm in women and ≥320 μm in men in the central subfield
* Lipid exudates involving the central subfield on spectral domain OCT.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

* Treatment for diabetic macular edema within the prior 4 months.
* Panretinal photocoagulation within the prior 4 months or anticipated need for panretinal photocoagulation within the next 6 months
* major ocular surgery within the prior 4 months
* myocardial infarction, other cardiac event requiring hospitalization, cerebrovascular accident, transient ischemic attack, or treatment for acute congestive heart failure occurred within 4 months before randomization
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an intrauterine device (IUD), or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - South Coast Retina Center; Carson, McBeath, Boswell, Inc, Huntington Beach, California
  - South Coast Retina Center; Carson, McBeath, and Boswell, Inc, Long Beach, California
  - Retina Partners, Santa Monica, California
  - South Coast Retina Center; Carson, McBeath, Boswell, Inc, Torrance, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.46) | 67 (8.83) | 65.75 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity as Measured by ETDRS at 6 and 12 Months
Description: Compare Group 1 and Group 2 for best correct visual acuity (BCVA), as assessed by the number of letters read correctly on the ETDRS eye chart at a starting test distance of 4 meters.
Time Frame: 6-12 months
Measure: Mean (Standard Deviation); unit: letters read correctly
Units Other Than Participants: Eyes
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
Number analyzed (Participants) | 12 | 12
Number analyzed (Eyes) | 12 | 12
letters read correctly
  6 Months | 78 (9.98) | 73.92 (8.40)
  12 Months | 77.92 (9.61) | 74.83 (8.32)

2. Secondary Outcome: Percentage of Eyes With Improvement of Lipid Deposits in the Central Subfield as Measured on OCT and Fundus Photography
Time Frame: 12 months
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 12 | 12
percentage of eyes | 70 | 83

3. Secondary Outcome: Percentage of Eyes With Complete Resolution of Lipid Deposits in the Central Subfield as Measured on OCT and Fundus Photography
Time Frame: 12 months
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 12 | 12
percentage of eyes | 60 | 58

4. Secondary Outcome: Number of Eyes With Complete Resolution in the Central Subfield as Measured on OCT and Fundus Photography
Time Frame: 12 months
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 12 | 12
eyes | 7 | 7

5. Secondary Outcome: Percentage of Eyes With Improvement in Lipid Deposits Throughout the Macular Grid as Measured by OCT and Fundus Photography
Time Frame: 12 months
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 12 | 12
percentage of eyes | 90 | 92

6. Secondary Outcome: Percentage of Patients With Complete Resolution of Lipid Deposits Throughout the Macular Grid as Measured on OCT and Fundus Photography
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

7. Secondary Outcome: Number of Eyes With Complete Resolution of Lipid Deposits Throughout the Macular Grid as Measured by OCT and Fundus Photography
Time Frame: 12 months
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 12 | 12
eyes | 0 | 0

8. Secondary Outcome: Incidence and Severity of Ocular Adverse Events as a Measure of Safety and Tolerability
Time Frame: 12 months
Population: eyes
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 4

9. Secondary Outcome: Incidence and Severity of Other Adverse Events as a Measure of Safety and Tolerability
Time Frame: 12 months
Population: eyes
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
Number analyzed (Participants) | 12 | 12
Participants | 9 | 9

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Diabetic Macular Edema Treatment Group (Group 1) | Diabetic Macular Edema and Lipid Treatment Group (Group 2)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/12 | 2/12
Other Adverse Events (participants affected / at risk) | 9/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetic Macular Edema Treatment Group (Group 1) (N=12) | Diabetic Macular Edema and Lipid Treatment Group (Group 2) (N=12)
Cysticercosis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Tapeworm - recovered with sequelae
Low Hemoglobin (Cardiac disorders) | 1 (1) | 0 (0) — low hemoglobin due to congestive heart failure
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Appendix Surgery (Infections and infestations) | 0 (0) | 1 (2)
Heart Attack (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetic Macular Edema Treatment Group (Group 1) (N=12) | Diabetic Macular Edema and Lipid Treatment Group (Group 2) (N=12)
Ear Infection (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Elevated Blood Pressure (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 3 (3)
Decreased Liver Function (Renal and urinary disorders) | 0 (0) | 1 (2)
Branch Retinal Artery Occlusion (Eye disorders) | 0 (0) | 1 (1)
Headache (Vascular disorders) | 1 (1) | 0 (0)
Shingles (Immune system disorders) | 1 (1) | 0 (0)
Elevated Triglycerides (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Central Retinal Vein Occlusion (Eye disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Ear Infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ocular Hypertension (Eye disorders) | 1 (1) | 0 (0)
Broken Wrist (Social circumstances) | 1 (1) | 0 (0)
Allergic conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Right Hip Injury (Social circumstances) | 1 (1) | 0 (0)
Drug Administration Error (Product Issues) | 1 (1) | 0 (0) — Incorrect drug administered
Subconjunctival Hemhorrage (Eye disorders) | 0 (0) | 1 (1)
Visual Acuity Loss (Eye disorders) | 1 (1) | 1 (1)
Metastatic Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Floater (Eye disorders) | 0 (0) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT02448446/Prot_SAP_000.pdf